CLINICAL TRIAL: NCT01104376
Title: Effect of Cytochrome P450 2B6 Genetic Polymorphism and Voriconazole on CYP2B6 Activity in Healthy Volunteers
Brief Title: Determine the Effects of Gene Differences and Voriconazole on Enzyme CYP2B6 Activity in the Liver in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Zeruesenay Desta, Associate Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0808-16; R01GM078501 (NIH)
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Efavirenz, Metabolism and Pharmacokinetics Changes
Keywords: Cytochrome P450; CYP2B6; Voriconazole; Efavirenz; Pharmacokinetics; Drug-Interactions; Pharmacogenetics; Healthy volunteers
MeSH Terms: interventions — efavirenz; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYP2B6 (Experimental): Healthy volunteers will receive Efavirenz and Vericonazole as follow:
  In phase 1 day 1 (control phase) a single 100mg dose of efavirenz will be administered. In phase 2 (voriconazole pretreatment phase), the subject will be pretreated with voriconazole (400mg twice daily on phase 2 day 8 and then 200mg twice daily for the next consecutive 8 days. In phase 3 (efavirenz plus voriconazole phase), the subject will receive on phase 3 day 10 100mg single dose of efavirenz along with 200mg of voriconazole twice daily.
  Interventions: Drug: Efavirenz; Drug: voriconazole

INTERVENTIONS:
Drug: Efavirenz — In phase 1 day 1 (control phase) a single 100mg dose of efavirenz will be administered.
  In phase 2 (voriconazole pretreatment phase), the subject will be pretreated with voriconazole (400mg twice daily on phase 2 day 8 and then 200mg twice daily for the next consecutive 8 days. In phase 3 (efavirenz plus voriconazole phase), the subject will receive on phase 3 day 10 100mg single dose of efavirenz along with 200mg of voriconazole twice daily.
  Other Names: Sustiva
Drug: voriconazole — In phase 1 day 1 (control phase) a single 100mg dose of efavirenz will be administered.
  In phase 2 (voriconazole pretreatment phase), the subject will be pretreated with voriconazole (400mg twice daily on phase 2 day 8 and then 200mg twice daily for the next consecutive 8 days. In phase 3 (efavirenz plus voriconazole phase), the subject will receive on phase 3 day 10 100mg single dose of efavirenz along with 200mg of voriconazole twice daily.
  Other Names: Vfend

SUMMARY:
The purpose of this study is to see if administration of medicines and genetic differences affects the activity of a liver enzyme called CYP2B6 in healthy volunteers.

DETAILED DESCRIPTION:
The investigators will test the hypothesis that CYP2B6 genetic variants that show effects in vitro also influence the in vivo activity of CYP2B6 and its responsiveness to metabolic inhibition, using the metabolism of efavirenz (100 mg dose) as a marker of activity. The metabolism and pharmacokinetics of efavirenz will be determined in a total of 60 healthy volunteers with CYP2B6*1/*1, CYP2B6*1*6 and CYP2B6*6*6 at baseline (control) and after pretreatment with voriconazole.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 55 years of age.
* Healthy individuals without any significant medical conditions as determined by a screening performed at University.
* Adherence to the study dietary and medication restrictions.
* Willingness to refrain from smoking or use of tobacco or marijuana one week before the start of the study and until completion of the study which will be a total of 17 days.
* Ability to commit the time requested for this study.

Exclusion Criteria:

* Underweight (weighs less than 50kg or 110lb) or over weight [body mass index (BMI) greater than 32].
* Drug or alcohol abuse (more than 3 alcoholic drinks per day on a regular basis).
* History of intolerance or allergic reaction (e.g. rash) to efavirenz and/or voriconazole.
* Significant health conditions such heart, gastrointestinal disorders, liver, or kidney diseases that may be exacerbated during the course of the study.
* History or current psychiatric illness (e.g. depression, anxiety, or nervousness).
* History or current eye sight disturbances (e.g. blurred vision).
* Serious infection within the last 2 weeks.
* Blood donation within the past two months.
* Screening results that do not fall in a healthy range.
* Regularly taking prescriptions (except hormonal agents, e.g. oral contraceptives), over-the-counter, herbal or dietary supplements, and alternative medications and are unable or unwilling to stop taking them one week before and during the study periods.
* Female with a positive pregnancy test.
* Female breastfeeding.
* Females of child-bearing potential who are unable or unwilling to either practice abstinence or use appropriate birth control up until the study completion, which will take a total of 17 days.
* Participation in a research study involving intensive blood sampling and/or have use study drugs in the last two months.
* Employed or student under supervision of any of the investigators of this study.
* Inability to state a good understanding of this study including risks and requirements, and inability to follow the rules of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeruesenay Desta, PhD, Principal Investigator — IU Department of Medicine/Division of Clinical Pharmacology
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Desta Z, Metzger IF, Thong N, Lu JB, Callaghan JT, Skaar TC, Flockhart DA, Galinsky RE. Inhibition of Cytochrome P450 2B6 Activity by Voriconazole Profiled Using Efavirenz Disposition in Healthy Volunteers. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6813-6822. doi: 10.1128/AAC.01000-16. Print 2016 Nov. PMID 27600044

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study is started with Consent and screening (Laboratory and medical).Therefore 89 subjects gave consents and where screened. Of those 61 fully completed all phase of the study while 15 partially completed. The 13 subjects gave their consent and were screened, but they did not take any intervention because of abnormal labs.
Groups:
- CYP2B6 Activity: CYP2B6 activity was measured using efavirenz metabolism and pharmacokinetics at baseline and after pretreatment with voriconazole.
  In phase 1 day 1 (control phase) a single 100mg dose of efavirenz will be administered.
  In phase 2 (voriconazole pretreatment phase), the subject will be pretreated with voriconazole (400mg twice daily on phase 2 day 8 and then 200mg twice daily for the next consecutive 8 days. In phase 3 (efavirenz plus voriconazole phase), the subject will receive on phase 3 day 10 100mg single dose of efavirenz along with 200mg of voriconazole twice daily.
Period: Overall Study
Arm/Group | CYP2B6 Activity
Started | 89
Completed | 61
Not Completed | 28
Not completed — Withdrawal by Subject | 15
Not completed — Consented but excluded after labs | 13

BASELINE CHARACTERISTICS:
Arm/Group | CYP2B6
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 33
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Measure Efavirenz Clearance
Description: Effect of steady-state voriconazole on efavirenz Clearance in healthy volunteers (n=61) administered a single 100 mg oral dose of efavirenz at baseline (control phase) and after treatment with voriconazole to steady-state.
Time Frame: Baseline, 30 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24h after efavirenz
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | CYP2B6
Number analyzed (Participants) | 61
ml/min/kg
  Control | 45.51 (18.3)
  Vericonazole | 20.03 (8.5)

ADVERSE EVENTS:
Arm/Group | CYP2B6
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No